CLINICAL TRIAL: NCT04473599
Title: Stay Well at Home: A Text-messaging Study to Improve Mood and Help Cope With Social Distancing
Brief Title: Stay Well at Home: a Text-messaging Study Social Distancing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020-04-13162
Record Dates: First submitted 2020-07-13; First posted 2020-07-16 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Depressive Symptoms; Anxiety; COVID-19
Keywords: Mobile health; Text-messaging; Covid-19; Mental health; Coping
MeSH Terms: conditions — Depression; Anxiety Disorders; COVID-19; Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants are randomized to receive messages according to a random schedule (within a mico-randomized trial), delivered via a reinforcement learning policy or a control with mood ratings only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Uniform Random (Active Comparator): Participants will receive supportive text-messages for a period of 2 months. These text-messages have two categories: behavioral activation (BA) and coping skills. In this arm, participants will receive one of these types of messages daily on a random schedule in random time periods throughout the day.
  Interventions: Behavioral: Uniform random message delivery
- Reinforcement Learning (Experimental): In this arm we will test a reinforcement learning (RL) algorithm with a learned decision mechanism for the timing and type of text-messages. The algorithm learns from previous data (which messages were sent, what was the participants' mood) to maximize an increase in participants' mood.
  Interventions: Behavioral: Reinforcement learning message delivery
- Mood ratings only (Active Comparator): In this arm, participants will monitor their mood and receive random feedback based on mood responses.
  Interventions: Behavioral: Mood ratings only

INTERVENTIONS:
Behavioral: Uniform random message delivery — In this arm, the categories and timings of text-messages will be delivered to participants using a random schedule
  Arms: Uniform Random
Behavioral: Reinforcement learning message delivery — In this arm, the categories and timings of text-messages will be chosen by a reinforcement learning algorithm
  Arms: Reinforcement Learning
Behavioral: Mood ratings only — In this arm, participants will monitor their mood daily and receive feedback on that mood randomly
  Arms: Mood ratings only

SUMMARY:
The investigators have developed supportive text-messages in English and Spanish to help people cope with the stress and anxiety of COVID-19 social distancing. The purpose of this study is to examine if automated text-messages will improve depression and anxiety symptoms and enhance positive mood.

Additionally, the investigators will compare the effectiveness of sending messages on a random schedule (using a micro-randomized trial design) or sent by a reinforcement learning policy on overall change in depression and anxiety symptoms and daily mood during the 8-week study.

DETAILED DESCRIPTION:
The investigators will send participants supportive text-messages for a period of 2 months. These text-messages will include tips about behavioral activation and coping skills to deal with worries and stress. The investigators generated a message bank balanced such that 50% of all messages are related to behavioral activation (BA) and 50% messages involve different coping skills. Participants will receive one of these messages per day between 9:00 am and 6:00 pm. Participants will also receive a message asking them to rate their mood on a scale of 1-9 once a day 3 hours after the BA or coping message.

Participants will be randomized to:

1. a uniform random messaging group (micro-randomized trial design).
2. a reinforcement learning group with a learned decision mechanism for the timing and type of text-message. The algorithm learns from previous data (which messages were sent, what was the participants' mood) to maximize an increase in participants mood. No other data are collected from participants' phones.

The investigators will compare the effect of sending text-messages by a random schedule, and text-messaging chosen by the RL algorithm. This allows to both evaluate the effect of the individual intervention components over time within a micro-randomized trial design, and assess the added value of using RL to adapt the messaging scheme.

The investigators hypothesize that:

* Participant will show improvements in depression, anxiety symptoms and mood during the 60 day study.
* The participants in the group receiving reinforcement learning will have a greater improvement in depressive symptoms, anxiety and positive mood during the study than participants in the micro-randomized group.
* The investigators will find differential effects on mood ratings for the two categories of messages

ELIGIBILITY:
Inclusion criteria:

* Over 18 years old
* Own a mobile phone
* Speak English or Spanish

Exclusion criteria:

* Not owning a mobile phone
* Under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2020-04-17 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Depression scores | Change from baseline to 8 week follow-up
  Patient Health Questionnaire 9 item (PHQ-9). The PHQ-9 has scores from 0 to 27. Higher scores mean a worse outcome.
Anxiety scores | Change from baseline to 8 week follow-up
  General Anxiety Disorder 7 item (GAD-7). The GAD-7 has scores from 0 to 21. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Self reported mood ratings | 8 weeks
  The self-reported mood rating 3 hours after receiving a message. The score is from 0-9. A higher mood rating indicates a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Aguilera, PhD, Principal Investigator — UC Berkeley
Locations (1):
- University of California Berkeley, Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlies the results reported in the articles will be made available to researchers on request after deidentification.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After publication of the data, no end date
Access Criteria: Anyone with a methodologically sound proposal.

REFERENCES:
- [Derived] Haro-Ramos AY, Rodriguez HP, Aguilera A. Effectiveness and implementation of a text messaging intervention to reduce depression and anxiety symptoms among Latinx and Non-Latinx white users during the COVID-19 pandemic. Behav Res Ther. 2023 Jun;165:104318. doi: 10.1016/j.brat.2023.104318. Epub 2023 Apr 16. PMID 37146444
- [Derived] Aguilera A, Hernandez-Ramos R, Haro-Ramos AY, Boone CE, Luo TC, Xu J, Chakraborty B, Karr C, Darrow S, Figueroa CA. A Text Messaging Intervention (StayWell at Home) to Counteract Depression and Anxiety During COVID-19 Social Distancing: Pre-Post Study. JMIR Ment Health. 2021 Nov 1;8(11):e25298. doi: 10.2196/25298. PMID 34543230
- [Derived] Figueroa CA, Hernandez-Ramos R, Boone CE, Gomez-Pathak L, Yip V, Luo T, Sierra V, Xu J, Chakraborty B, Darrow S, Aguilera A. A Text Messaging Intervention for Coping With Social Distancing During COVID-19 (StayWell at Home): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2021 Jan 14;10(1):e23592. doi: 10.2196/23592. PMID 33370721